CLINICAL TRIAL: NCT03182270
Title: Clinical Evaluation Of Needle-based Confocal Laser Endomicroscopy in Cystic Tumors of the Pancreas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZS-1265
Record Dates: First submitted 2017-05-19; First posted 2017-06-09 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Cystic Tumors of Pancreas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pancreatic cysts (Experimental)
  Interventions: Diagnostic Test: nCLE

INTERVENTIONS:
Diagnostic Test: nCLE — Procedure: EUS-FNA Device: nCLE

SUMMARY:
This study focuses on pancreatic cysts, especially malignant pancreatic cysts. The primary hypothesis of the study is that using nCLE in addition to EUS-FNA and tissue sampling allows better characterization of pancreatic cysts and improves appropriate therapeutic decision-making. For physicians, integrating nCLE into the diagnostic algorithm of pancreatic cysts could impact patient management by: Ruling out malignancy for patients with benign appearing nCLE images. Characterizing more malignant tumors in the pancreas.

DETAILED DESCRIPTION:
1. Medical background: Pancreatic cysts are quite rare, but are being increasingly recognized due to the expanding use of cross-sectional imaging. They are classified into three main classes: pseudocysts, serous cysts and mucinous cystic neoplasms. Either intraductal papillary mucinous neoplasm (IPMN) or mucinous cyst adenomas / mucinous cystadenocarcinoma(MCN) Mucinous cystic neoplasms are considered to be malignant or pre-malignant and are considered for surgical resection, whereas pseudocysts and serous cysts are considered benign and with a low potential for malignancy. Pseudocysts and serous cysts are usually only considered for surgical resection when symptomatic or enlarging.
2. Clinical background:

   2.1. Endoscopic Ultrasound (EUS) is the diagnostic method of choice when a pancreatic lesion is found incidentally on cross-sectional imaging. Endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) is a procedure where a target tissue in proximity to the GI tract is biopsied using a fine needle guided in real time by an ultrasound probe fixed at the tip of an endoscope. It may therefore be applied to pancreatic lesions, or lymph nodes examination.

   2.2. The principle of needle-based Confocal Laser Endomicroscopy (nCLE) is to image organs within or adjacent to the GI tracts with a miniprobe inserted through an endoscopic needle. The fundamental technology as well as the principle of operation of nCLE are substantially similar to pCLE.
3. Clinical evidence: Previous studies enabled to define interpretation criteria on the micro-structure of benign pancreatic cysts. Less data is available on malignant pancreatic cysts, except for a few images done in a pilot study of identification of pancreatic cystic neoplasms.
4. Objectives:

   4.1 The primary objective of the study is to assess the diagnostic performance of the Cellvizio nCLE system in diagnosing pancreatic cysts, when associated with other diagnostic information.

   4.2 The secondary objectives are to assess the potential impact of the Cellvizio nCLE system on patient management and validate the interpretation classification criteria that were created during the previous studies.
5. Design:

This study will be conducted in a single center in China.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years of age.
* Patient indicated for a first EUS-FNA for a pancreatic cyst or
* Patients who had previous non-diagnostic tissue sampling taken during a previous EUS-FNA for pancreatic cyst more than three months ago.
* Patient with known pancreatic cyst detected at cross-sectional imaging
* Willing and able to comply with study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

* Subjects for whom EUS-FNA procedures are contraindicated
* Known allergy to fluorescein dye
* If female, pregnant based on a positive hCG serum or an in vitro diagnostic test result or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of the Cellvizio nCLE system in the characterization of pancreatic cysts | Within 6 months after the end of Follow-up period
  Diagnostic performance of the Cellvizio nCLE system compared with pathological results or consensus review at a multidisciplinary tumor board meeting

SECONDARY OUTCOMES:
Safety data on nCLE during EUS-FNA procedure (rate of procedure related complication) | Within 3 months after the end of the enrollment period
  The rate of procedure related complication including bleeding, post-procedure pancreatitis and perforation
Feasibility data on nCLE during EUS-FNA procedure (rate of successful nCLE procedure) | Within 3 months after the end of the enrollment period
  The rate of successful nCLE procedure

CONTACTS AND LOCATIONS:
Overall Officials: Aiming Yang, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided